CLINICAL TRIAL: NCT04426175
Title: Precision of 2D vs 3D Low Energy Femto-LASIK: Intraoperative and Postoperative OCT-based Study
Brief Title: Z8 OCT-controlled 2D vs 3D LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zentrumsehstarke Hamburg (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPFEM-0007-DE
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Myopia; Astigmatism
Keywords: Femtosecond Laser Assisted Laser in Situ Keratomileusis; LASIK; FEMTO LDV Z8
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2D LASIK (Experimental): With the 2D method, the flap resection is created in a planar mode (xy-plane), without vertical cut, at the requested depth.
  Interventions: Device: 2D and 3D cutting method using a low energy Femtosecond laser LDV Z8 for LASIK flap cutting
- 3D LASIK (Experimental): With the 3D method, the flap resection is done in a three-dimensional mode, at the requested depth, with the requested diameter and the desired border (side cut) angle
  Interventions: Device: 2D and 3D cutting method using a low energy Femtosecond laser LDV Z8 for LASIK flap cutting

INTERVENTIONS:
Device: 2D and 3D cutting method using a low energy Femtosecond laser LDV Z8 for LASIK flap cutting — 2D and 3D cutting methods were randomly used in same subjects

SUMMARY:
The aim of this study was to test the hypothesis that OCT-guided 110 µm targeted flaps will result in accurate, predictable, and precise thickness flaps, with low complication rates when performed and compared using both 2D and 3D flap geometry applications and how it correlated to visual experience and quality of life responses during the early postoperative period.

DETAILED DESCRIPTION:
It has been postulated that it is possible with the Ziemer Femtosecond LDV laser system to create reproducible flaps in terms of thickness and predictability. The aim of this study was to test the hypothesis that OCT-guided 110 µm targeted flaps will result in accurate, predictable, and precise thickness flaps, with low complication rates when performed and compared using both 2D and 3D flap geometry applications. Patient-reported outcomes are increasingly incorporated into clinical trials as they provide access to valuable information on the physical experience of the patient during and after the treatment. A questionnaire will therefore also be introduced in this study to evaluate how well self-reported pain, visual experience, and quality of life responses are correlated with flap geometries in both groups during the early postoperative period. The study holds direct medical benefit to the patient in this that they received an immediate improvement in his/her unaided vision. Moreover, the patient's participation contributes to the medical knowledge about the use of femtosecond lasers for refractive surgery, in particular in view of the use of intraoperative OCT visualization tools. The patients will gain access to the newest technology available for refractive surgery namely a low pulse energy high-frequency femtosecond laser.

ELIGIBILITY:
Inclusion Criteria:

Key inclusion criteria as described by the German Commission for Refractive Surgery (KRC) are:

* The recommended range of application for the correction of myopia is up to -8.00 D and for the correction of astigmatism up to 5.00 D.
* The limited for LASIK correction of myopia is up to -10.00 D and correction of astigmatism up to 6.00 D. If myopic astigmatism is to be corrected, the values for myopia and astigmatism must be added together.
* The recommended range for correction of hyperopia is up to 3.00 D. Up to 4.00 D is the range of limited application for hyperopia.
* Age ≥18 years with stable eyesight for over 12 months.

Exclusion Criteria:

Key exclusion criteria as described by the German Commission for Refractive Surgery (KRC):

* preoperative corneal thickness less than 480 μm
* predicted stromal thickness under the flap after ablation of less than 250 μm
* chronic progressive corneal disease and forme fruste keratoconus
* surgery before the age of 18 years
* symptomatic cataract
* Glaucoma with a marked loss of visual field
* Exudative macular degeneration.
* Concurrent participation in another ophthalmological clinical study

Exclusion criteria irrespective of the KRC criteria:

* Undergone former eye surgery
* Contact lens wear within the two weeks prior to commencement of preoperative measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-04-23 (Actual); Study Completion 2020-04-23 (Actual)

PRIMARY OUTCOMES:
Predictability of central flap thickness in OCT-controlled 110 µm LASIK | 1 month postoperatively
  Analyze central flap thickness in OCT-controlled 110 µm LASIK and to report on intended versus achieved flap thickness of one group with a 2D flap geometry in one eye and another group with a 3D flap geometry in the contralateral eye. All OCT measurements will be done in micron metres (µm).

SECONDARY OUTCOMES:
Comparison of intraoperative flap thickness with pre- and postoperative results | 1 week, 1 month
  Measurement of corneal thickness pre flap creation (Corneal Pachymetry measurements expressed in µm indicate the thickness of the cornea before flap was created. This measurement will serve as the baseline measurement. Pachymetry measured again after the flap was created and lifted by means of optical and ultrasonic pachymetry(µm) for both groups and to be compare with postoperative AS-OCT measurements also measured in µm.This will indicate how accurate the intraoperative flap thickness compare to the 1 week and 1 month thickness measurements as swelling and inflammatory processes could influence postoperative measurements.
Postoperative planarity | 1 week, 1 month
  Assessment of several measurements taken along the corneal cut on superior, nasal, inferior and temporal points in order to compare the uniformity of the cut between 2D vs 3D geometries. Measurments will be done by means of AS-OCT,measured in µm units.Measurements at two different follow up periods will be analyzed and compared in order to rule out the role that inflammation could possibly play.
Intraoperative flap morphology | During surgery
  Observations that are defined by different scales in order to report on important features pertaining to 2D and 3D intraoperative flap geometries eg. the presence and extent of opaque bubble layer (OBL), ease of flap lifting and stromal bed quality in both groups . Intraoperative flap morphology assessment to be done as soon as the flap was created in terms of presence of an opaque bubble layer (no OBL, 30-40% of flap surface, >40% of flap surface). Once the flap was lifted to report on ease of flap lifting (easy/sticky/can not lift) and to describe the stromal bed quality (smooth,tissue bridges, rastered, lines).
Postoperative flap properties | 1 week, 1 month
  Evaluate flap properties by means of slit lamp biomicroscopy examination. The flap's visual appearance seen with the slit lamp to be described and documented as per the suggested scales during 2 specified follow up visits in terms of edge quality and visibility ('yes/no' If yes= extreme fine line, distinct line or irregular edge), border shape (round, irregular) and interface quality (smooth, lines, cobblestones, grids, microstriae) and be compared between flap geometries (2D and 3D flaps).
Visual outcomes | 1 day, 1 week, 1 month
  Compare pre- and postoperative visual acuity (UDVA, CDVA) measurements by means of a Snellen Visual Acuity chart and be expressed in decimal that will be converted to logMar units for the purpose of statistical analysis.
Patient reported Outcomes: early recovery period | 1 day, 2Day, 1 week follow up
  Conduct a non validated Patient Reported Outcome (PRO) questionnaire adopted and based on the 'Brief Pain Inventory' questionnaire [Porela-Tiihonen] to assess patient's early visual perceptions and pain experience related to their own functional status and wellbeing and to compare between the two eyes since each undergone different cutting geometry (2D vs 3D) methods.
Complications | Intra- and postoperatively up to 1 month follow up
  Report and document any intra- and postoperative complications that may occur during the time of the procedure or at the 1 month follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Linke, MD, Principal Investigator — Zentrumsehstarke Hamburg
Locations (1):
- Zentrumsehstärke, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
It is not clear yet to what extend IPD will be implemented. Patient privacy and confidentiality are the most important factors to consider. We consider sharing limited information upon request.

REFERENCES:
- [Background] Huhtala A, Pietila J, Makinen P, Uusitalo H. Femtosecond lasers for laser in situ keratomileusis: a systematic review and meta-analysis. Clin Ophthalmol. 2016 Mar 7;10:393-404. doi: 10.2147/OPTH.S99394. eCollection 2016. PMID 27022236
- [Background] Eldaly ZH, Abdelsalam MA, Hussein MS, Nassr MA. Comparison of Laser In Situ Keratomileusis Flap Morphology and Predictability by WaveLight FS200 Femtosecond Laser and Moria Microkeratome: An Anterior Segment Optical Coherence Tomography Study. Korean J Ophthalmol. 2019 Apr;33(2):113-121. doi: 10.3341/kjo.2018.0035. PMID 30977320
- [Background] Pajic B, Vastardis I, Pajic-Eggspuehler B, Gatzioufas Z, Hafezi F. Femtosecond laser versus mechanical microkeratome-assisted flap creation for LASIK: a prospective, randomized, paired-eye study. Clin Ophthalmol. 2014 Sep 22;8:1883-9. doi: 10.2147/OPTH.S68124. eCollection 2014. PMID 25284975
- [Background] Tomita M, Chiba A, Matsuda J, Nawa Y. Evaluation of LASIK treatment with the Femto LDV in patients with corneal opacity. J Refract Surg. 2012 Jan;28(1):25-30. doi: 10.3928/1081597X-20111213-01. Epub 2011 Dec 19. PMID 22185466
- [Background] Pietila J, Huhtala A, Makinen P, Uusitalo H. Flap characteristics, predictability, and safety of the Ziemer FEMTO LDV femtosecond laser with the disposable suction ring for LASIK. Eye (Lond). 2014 Jan;28(1):66-71. doi: 10.1038/eye.2013.244. Epub 2013 Nov 15. PMID 24232315
- [Background] Pietila J, Huhtala A, Makinen P, Salmenhaara K, Uusitalo H. Laser-assisted in situ keratomileusis flap creation with the three-dimensional, transportable Ziemer FEMTO LDV model Z6 I femtosecond laser. Acta Ophthalmol. 2014 Nov;92(7):650-5. doi: 10.1111/aos.12333. Epub 2013 Dec 26. PMID 24373615
- [Background] Porela-Tiihonen S, Kaarniranta K, Kokki M, Purhonen S, Kokki H. A prospective study on postoperative pain after cataract surgery. Clin Ophthalmol. 2013;7:1429-35. doi: 10.2147/OPTH.S47576. Epub 2013 Jul 15. PMID 23885165